CLINICAL TRIAL: NCT02405923
Title: Clinical Trial Evaluating the Effects on Growth, Safety and Tolerance of a Rice Protein Hydrolysate Formula Compared to a Cow's Milk Extensively Hydrolysed Protein Formula in Infants With Cow's Milk Protein Allergy
Brief Title: Growth, Safety and Tolerance of a Rice Protein Hydrolysate Formula in Infants With Cow's Milk Protein Allergy
Acronym: GRITO-14
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment longer than expected and without the expected success
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRITO-14
Record Dates: First submitted 2014-11-13; First posted 2015-04-01 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HRF (Rice formula) (Experimental): Hydrolyzed Rice Protein Formula (HRF)
  Interventions: Other: HRF
- eHF (Extensive Hydrolysed Formula) (Placebo Comparator): Extensive Hydrolysed Cow's Milk Protein Formula (eHF)
  Interventions: Other: eHF

INTERVENTIONS:
Other: HRF — The subject will take the formula for a period of 12 months.
  Other Names: HRF-1 from 0 to 6 months of age; HRF-2 from 6 months of age onwards
  Arms: HRF (Rice formula)
Other: eHF — The subject will take the formula for a period of 12 months.
  Other Names: eHF-1 from 0 to 6 months of age; eHF-2 from 6 months of age onwards
  Arms: eHF (Extensive Hydrolysed Formula)

SUMMARY:
This is a multicenter, controlled, randomized, prospective, non-inferiority, double blind intervention trial to evaluate the children growth (at 6, 9 and 12 months) using a rice hydrolysed protein formula compared to an extensively cow's milk protein hydrolysed formula for the management of Cow's Milk Protein Allergy (CMPA).

DETAILED DESCRIPTION:
The main purpose of this study is to demonstrate that the rice protein hydrolysed based formula manufactured by Ordesa ensures proper growth and as secondary outcomes, that the formula is devoid of any risk of arsenic or other potential contaminants toxicity and its effect on the duration of CMA (Cow Milk Allergy) from cow's milk protein allergy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects up to 10 months old with clinical history of a reaction to cow's milk protein and/or confirmed diagnosis (up to grade II anaphylaxis) of allergy to cow's milk protein by one of the following criteria, within two months prior to the baseline visit are eligible to enter the study:

  * Negative or positive skin prick tests ( fresh milk, rice, casein hydrolysates)
  * Negative or positive specific IgE for cow's milk proteins (alphalactalbumine, betalactoglobuline, caseine and cow's milk)
  * Negative or positive Milk Atopy Patch Test
  * Positive Double Blind Placebo Control Food Challenge (DBPCFC) with cow milk
* Gestational Age 37-42 weeks inclusive
* Apgar SCORE >7 at 5 minutes
* Singleton birth
* Birth weight ≥2.500 g
* Written informed consent

Exclusion Criteria:

* Previous signs of allergy to any extensively hydrolysed formula
* Confirmed history of acute severe, potentially life threatening reaction after isolated accidental ingestion of cow's milk e.g. history of anaphylactic reaction, graded more or equal to grade III, as this could not be compatible with an allocation to the eHF group
* Daily formula intake < 100 ml
* Major congenital malformations or neonatal diseases
* Severe concurrent or chronic diseases
* Intrauterine growth retardation
* Neonatal infections ( e.g. CMV, HIV)
* Simultaneous participation in other clinical trials
* Parents not signing written informed consent
* Unable to adhere to protocol requirements or study visits due to non compliance of parents or caregivers.
* Liver, kidney, haematological abnormalities as judged clinically by investigators at baseline.

Max Age: 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Growing change | 6 months
  To evaluate the children growth using a rice hydrolysed protein formula compared to an extensively cow's milk protein hydrolysed formula for the management of CMPA.

SECONDARY OUTCOMES:
Nutritional adequacy | 6 months
  To monitor nutritional adequacy in terms of anthropometrics and proteic status.
Contaminants | 6 months
  To monitor the presence of possible contaminants in urine and hair samples coming from both infant formula groups (only in children exclusively or predominantly formula fed; ideally recruited from 0 to 6 months). Moreover the presence of possible contaminants will be evaluated also in powder formula and formula from baby bottles (only in 12 patients, randomly chosen).
Tolerance acquisition to cow's milk protein measured by a cow milk OFC (Open Food Challenge) | 6 months
  To evaluate the acquisition of tolerance between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Mireia, MD, Principal Investigator — Laboratorios Ordesa
Locations (5):
- France (2):
  - Hôpital Necker-Enfants Malades, Paris, Cedex 14
  - Hôpital Saint Vincent-de-Paul, Lille, Lille Cedex
- Spain (3):
  - Hospital Infantil Virgen del Rocío, Seville, Andalusia
  - Hospital Materno Infantil de Málaga, Málaga
  - Hospital Universitari i Politècnic La Fe, Valencia